CLINICAL TRIAL: NCT01381016
Title: Estrogen Sensitivity and Ovulatory Dysfunction in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-0293
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Obesity; Infertility
Keywords: LH pulsatility; Obesity; Reproduction
MeSH Terms: conditions — Obesity; Infertility | interventions — Estradiol; Gonadotropin-Releasing Hormone; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Normal Weight (Other): Group 1: Normal weight (BMI 18-25 kg/m2)
  Subjects were instructed to apply 0.1 mg/d transdermal estrogen (Estradiol) for one month. Pituitary response was assessed to determine how estradiol administration altered pituitary sensitivity to Gonadotropin-releasing hormone - GnRH. Subjects who failed to initiate a menstrual period following 40 days on the patch were instructed to take 200 mg daily of progesterone for 10 days or as long as deemed necessary.
  Interventions: Drug: Estradiol; Drug: Gonadotropin-releasing hormone (GnRH); Drug: Progesterone
- Group 2 - Obese (Experimental): Group 2: Obese (BMI >30 kg/m2)
  Subjects were instructed to apply 0.1 mg/d transdermal estrogen (Estradiol) for one month. Pituitary response was assessed to determine how estradiol administration altered pituitary sensitivity to Gonadotropin-releasing hormone - GnRH. Subjects who failed to initiate a menstrual period following 40 days on the patch were instructed to take 200 mg daily of progesterone for 10 days or as long as deemed necessary.
  Interventions: Drug: Estradiol; Drug: Gonadotropin-releasing hormone (GnRH); Drug: Progesterone

INTERVENTIONS:
Drug: Estradiol — Subjects were instructed to apply 0.1 mg/d transdermal estrogen for one month.
  Other Names: Climara, transdermal estrogen
Drug: Gonadotropin-releasing hormone (GnRH) — Pituitary response was assessed to determine how estradiol administration alters pituitary sensitivity to GnRH.
  Other Names: Lutrelef or gonadorelin acetate
Drug: Progesterone — Subjects who failed to initiate a menstrual period following 40 days on the patch were instructed to take 200 mg daily of progesterone for 10 days or as long as deemed necessary.
  Other Names: Prometrium or medroxyproge sterone acetate

SUMMARY:
The sole purpose of this study is to evaluate pathophysiology of disease. The disease state that is being evaluated is the obesity-related alterations in reproductive hormones

* The obesity epidemic in the United States is advancing at an accelerated pace. It is estimated that by 2015, 41% of U.S. adults will be obese as defined by a body mass index (BMI) of greater than 30 kg/m2. The U.S. government's 2010 Dietary Guidelines regard obesity as the single greatest health hazard in this century. Female adult obesity is associated with menstrual cycle irregularities, ovulatory dysfunction and a higher risk of obstetrical complications. This reproductive phenotype of obesity is worsened by further increases in BMI and is not solely due to anovulatory infertility. While the association of adiposity with subfertility is well documented in population studies, the underlying mechanisms remain poorly understood. The main objective of this proposal is to clarify the nature of the obesity-related reproductive endocrine abnormalities and identify potential etiologies amenable to therapy.
* Hypothesis: The hypothalamic-pituitary axis is abnormally sensitive to estradiol negative feedback in obesity.

DETAILED DESCRIPTION:
* Design: paired assessments Pre and Post estrogen administration in obese and normal weight women
* AIM 1: To test the pituitary and hypothalamic responsiveness in obesity, we will examine the luteinizing hormone (LH) and follicle-stimulating hormone (FSH) pulsatility during frequent blood sampling.
* AIM 2: To test the ovarian responsiveness in obesity, we will examine urinary reproductive hormones (E1c, estrone conjugates, and Pdg, pregnanediol glucuronide) over an entire menstrual cycle.
* AIM 3: To test the hypothesis that central adiposity is associated with reproductive hormone alterations in obesity, we will quantitatively assess body composition by dual energy x-ray absorptiometry (DXA).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-42 at study entry
* Regular menstrual cycles every 25-40 days
* BMI 18- 25 kg/m2 or ≥30kg/m2
* Good general health
* Prolactin and thyroid-stimulating hormone (TSH) within normal laboratory ranges at screening
* Baseline hemoglobin >11 gm/dl.

Exclusion Criteria:

* Positive screen for Activated Protein C resistance
* Any contraindications to exogenous estrogen, including previous thromboembolic events or stroke, history of an estrogen-dependent tumor, active liver disease, undiagnosed abnormal uterine bleeding, hypertriglyceridemia, smoking, hypertension
* History of chronic disease affecting hormone production, metabolism or clearance (including diabetes mellitus) or abnormal renal or liver function at screening, such as elevated aspartate or alanine aminotransferases or elevated blood urea nitrogen (BUN) or creatinine
* Current use of thiazolidinediones or metformin (known to interact with reproductive hormones)
* Use of hormones affecting hypothalamic-pituitary ovarian axis within three months of enrollment
* Strenuous exercise (>4 hours per week)
* Pregnancy, breast-feeding or current active attempts to conceive

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Polotsky, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Background] Jain A, Polotsky AJ, Rochester D, Berga SL, Loucks T, Zeitlian G, Gibbs K, Polotsky HN, Feng S, Isaac B, Santoro N. Pulsatile luteinizing hormone amplitude and progesterone metabolite excretion are reduced in obese women. J Clin Endocrinol Metab. 2007 Jul;92(7):2468-73. doi: 10.1210/jc.2006-2274. Epub 2007 Apr 17. PMID 17440019
- [Background] Rochester D, Jain A, Polotsky AJ, Polotsky H, Gibbs K, Isaac B, Zeitlian G, Hickmon C, Feng S, Santoro N. Partial recovery of luteal function after bariatric surgery in obese women. Fertil Steril. 2009 Oct;92(4):1410-1415. doi: 10.1016/j.fertnstert.2008.08.025. Epub 2008 Sep 30. PMID 18829008
- [Derived] Roth LW, Allshouse AA, Lesh J, Polotsky AJ, Santoro N. The correlation between self-reported and measured height, weight, and BMI in reproductive age women. Maturitas. 2013 Oct;76(2):185-8. doi: 10.1016/j.maturitas.2013.07.010. Epub 2013 Aug 16. PMID 23958434

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Group 1 "Control": Normal weight (BMI 18-25 kg/m2)
  Estradiol, Lutrelef or gonadorelin
- Experimental: Group 2 "Experimental": Obese (BMI >30 kg/m2)
  Estradiol, Lutrelef or gonadorelin
Period: Overall Study
Arm/Group | Control | Experimental
Started | 13 | 17
Completed | 10 | 11
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Screen Failure | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 17 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 29 [23 to 41] | 31.76 [19 to 39] | 30.57 [19 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: Luteinizing Hormone Pulse Amplitude
Description: The study is powered on luteinizing hormone pulse amplitude because it is the clinical outcome for which the most data is available. The primary comparison is whether there is a significant reduction in the pulse amplitude in the obese between the pre- and post-treatment periods and whether there is no change in the pulse amplitude in the normal weight patients between the pre and post-treatment periods.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: IU/L
Groups:
- Group 1 - Normal Weight: Group 1: Normal weight (BMI 18-25 kg/m2)
  Estradiol, Lutrelef or gonadorelin
- Group 2 - Obese: Group 2: Obese (BMI >30 kg/m2)
  Estradiol, Lutrelef or gonadorelin
Arm/Group | Group 1 - Normal Weight | Group 2 - Obese
Number analyzed (Participants) | 10 | 11
IU/L | 2.73 (.46) | 1.12 (.19)

2. Primary Outcome: Luteinizing Hormone Pulse Amplitude
Time Frame: Post estradiol at one month
Measure: Mean (Standard Error); unit: IU/L
Groups:
- Control: Group 1: Normal weight (BMI 18-25 kg/m2)
  Estradiol, Lutrelef or gonadorelin
- Experimental: Group 2: Obese (BMI >30 kg/m2)
  Estradiol, Lutrelef or gonadorelin
Arm/Group | Control | Experimental
Number analyzed (Participants) | 10 | 11
IU/L | 2.18 (.4) | 1.59 (.29)

ADVERSE EVENTS:
Description: 2/13 subjects enrolled as controls were considered screen failures, thus only 11 subjects were considered participants "at risk" in the control group.
  2/17 subjects enrolled in experimental group were considered screen failures, thus only 15 subjects were considered participants "at risk" in the experimental group.
Arm/Group | Control | Experimental
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/15
Other Adverse Events (participants affected / at risk) | 0/11 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=11) | Experimental (N=15)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No